CLINICAL TRIAL: NCT03588546
Title: FASENRA Subcutaneous Injection 30 mg Syringe Specific Clinical Experience Investigation for Long-term Use
Brief Title: FASENRA SCEI for Long-term Use
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250C00057
Record Dates: First submitted 2018-05-25; First posted 2018-07-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Fasenra Benralizumab Bronchial asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
The purpose of the investigation is to confirm the safety and efficacy under the post-marketing actual long-term use of FASENRA Subcutaneous Injection 30 mg Syringe.

DETAILED DESCRIPTION:
The purpose of the investigation is to confirm the followings under the post-marketing actual long-term use of FASENRA Subcutaneous Injection 30 mg Syringe.

1. Detection of unexpected Adverse Drug Reactions
2. To grasp development of Adverse Drug Reactions
3. To grasp contributing factors possibly having an impact on the safety and efficacy
4. Development of key investigational safety specification (serious infection).

ELIGIBILITY:
Inclusion Criteria:

-The evaluable patients treated with Fasenra for the first time due to "Bronchial asthma (only the patients with intractable bronchial asthma which could not be controlled with the existing therapy).

Exclusion Criteria:

-No past history of hypersensitivity to the components of Fasenra.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients treated with Fasenra for the first time due to "Bronchial asthma (only the patients with intractable bronchial asthma which could not be controlled with the existing therapy).
Sampling Method: Non-Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Incidences of adverse drug reactions (ADRs) [all ADRS, unexpected ADRs and key investigational safety specification (serious infection)] | 1 year

SECONDARY OUTCOMES:
Change scores from baseline in Asthma Control Questionnaire (ACQ) with exploring a factor to affect them by patient's background and treatment condition | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (29):
- Japan (29):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukuoka
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Yamagata
  - Research Site, Yamaguchi

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00057&attachmentIdentifier=e4c2acde-e375-4de3-91f5-199e6a0fab44&fileName=Clinical_Study_Report_(CSR)_Synopsis,_RIMS_FSN_D3250C00057.pdf&versionIdentifier=